CLINICAL TRIAL: NCT04310449
Title: Hard and Soft Tissue Alterations on the Use of Dual Zone Concept Versus Connective Tissue Graft At Flapless Maxillary Immediate Implant Placement. a 1-year Randomized Clinical Trial and Volumetric Study.
Brief Title: Volumetric Changes of Labial Soft Tissue Contour Following Different Approaches with Immediate Implant Placement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Misr International University (Other)
Responsible Party: Principal Investigator, Ahmed Abo El Futtouh, Clinical Director of Implant Program - Periodontology and Implantology Consultant, Misr International University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PER8273002
Record Dates: First submitted 2020-03-09; First posted 2020-03-17 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Dental Implant Placement
Keywords: Immediate implant placement; Connective tissue graft; dual-zone therapeutic concept; customized healing abutment; buccal soft tissue contour; volumetric analysis

STUDY DESIGN:
Intervention Model Description: • To compare the volumetric changes in the buccal soft tissue contour between immediate implants with CTG and customized healing abutments, and immediate implants with bone grafting in the dual zone and customized healing abutmnets
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dual zone concept and customized healing abutment (Experimental): Immediate implant placement with bone grafts in the dual zone and customized healing abutment.
  Interventions: Procedure: Dual zone concept and customized healing abutment
- Connective tissue graft and customized healing abutment (Active Comparator): immediate implant placement with CTG and customized healing abutment
  Interventions: Procedure: Connective tissue graft and customized healing abutment

INTERVENTIONS:
Procedure: Connective tissue graft and customized healing abutment — Immediate implant placement without flap raising using standard implant system protocol preparation will take place. Connective tissue grafts from the hard palate will be placed at the implant sites in a supraperiosteal partial dissection prepared at the buccal aspect. Sutures will be used to stabilize the graft, followed by customized healing abutment. Flowable composite will be injected at the gingival margin level to adapt to the sandblasted abutment, taking the shape of the socket at the marginal gingiva. Buccal groove will be made after the polymerization of this material for easier application. The abutments will be removed for final configurations of the apical part mimicking the emergence profile of the extracted tooth and finishing with laboratory discs and burs. The custom healing screw will be screwed to the implant.
  Other Names: zimmer biomed dental implants and connective tissue grafts and customized healing abutments
  Arms: Connective tissue graft and customized healing abutment
Procedure: Dual zone concept and customized healing abutment — Immediate implant placement without flap raising using standard implant system protocol preparation will take place. Followed by bone grafting following dual zone concept and customized healing abutment.
  Other Names: zimmer biomed dental implants and dual zone bone grafting and customized healing abutments
  Arms: Dual zone concept and customized healing abutment

SUMMARY:
Statement of the problem: Tooth extraction is followed by ridge alteration and soft tissue contour collapse. Different strategies were proposed to limit this collapse however, the ability of these techniques to mimic the original soft tissue contour and to maintain long term stability is unclear. Purpose : The aim of this study is to evaluate the volumetric difference of buccal soft tissue contour as well as the radiographic changes, following tooth extraction and immediate implant placement with dual zone concept versus connective tissue graft. Materials and Methods: Thirty patients with single maxillary anterior or premolar tooth indicated for extraction will participate in this study, 15 patient in each group. Group 1 (test group) will be treated by immediate implant placement (IIP) with particulate bone grafts in the dual zone (the bone zone and the tissue zone) and customized healing abutment. Group 2 (control group) IIP with connective tissue graft (CTG) and customized healing abutment. Patient allocation is random for the 2 groups. Data will be collected pre-surgically and at follow up periods (3,6,9&12 months and 6 months after delivery). Extra-oral scanning of the labial contour will be carried out to evaluate difference in contour gained and will be compared to the original contour and between treatment groups. Radiographic evaluation will be done using CBCT pre-operatively and at 12 months.

DETAILED DESCRIPTION:
After administration of local anaesthesia, the tooth will be extracted by the principle investigator without raising flaps, as atraumatically as possible by using periotomes without disturbing the papillary tissues (minimal traumatic extraction technique). After the extraction of the tooth, the socket will be carefully cleaned to excavate the granulation tissue in the marginal and apical regions. The allocation will be revealed to the principle investigator for the 3 implant groups after implant placement.

Group 1: extraction will occur and then followed by immediate implant placement,using standard implant system protocol preparation of the osteotomy will take place. Initial drill will be placed palatally till final drill reached. Placement of the implant without any raising of the flap will be performed in the correct implant position. Primary stability of the implant will be measured by rotational insertion torque value, to be ≥30Ncm (37). Particulate bone grafts are packed in the gap between the implant and the buccal plate of bone and the tissue (dual zone), Followed by customized healing abutment, the temporary cylindrical abutment twill be screwed to the implant and then flowable composite will be injected at the gingival margin level to adapt to the abutment that will be sand-blasted previously for mechanical retention of the composite, taking the shape of the socket at the marginal gingiva, but will only seal the socket without extending deeper apically in the soft tissue. A buccal groove will be made after the polymerization of this material for easier application. The abutments will be removed for final configurations of the apical part mimicking the emergence profile of the extracted tooth and finishing with laboratory discs and burs. The custom healing screw will then be screwed to the implant with the correct torque.

Group 2: Tooth extraction and immediate implant placement as mentioned. Connective tissue grafts will be harvested from the hard palate and placed at the implant sites in a supraperiosteal partial dissection (pouch technique) prepared at the buccal aspect without using vertical incisions and without flap elevation. Sutures will be used to stabilize the graft in its desired place, then will be covered by a customized healing abutment that will be done as mentioned before.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have at least one non-restorable maxillary anterior or premolar tooth with sound adjacent teeth.
2. Adults at or above the age of 18.
3. Intact thick biotype gingival tissue with at least 2mm band of keratinized tissue.
4. Buccal bone thickness should be 1mm or less assessed in CBCT with good apical bone.
5. Sagittal root position type 1 as described by Kan et al(30).
6. Good oral hygiene
7. Patient accepts to provide an informed consent.

Exclusion Criteria:

1. Smokers
2. Pregnant and lactating females.
3. Medically compromised patients. , as Uncontrolled diabetic patients, patients taking bisphosphonates injection for treatment of osteoporosis, patients with active cardiac diseases, patients undergoing radiotherapy or chemotherapy, or any other medical and general contraindications for the surgical procedure (i.e. ASA score ≥III) (31)
4. Patients with active infection related at the site of implant/bone graft placement.
5. Patients with untreated active periodontal diseases.
6. Patients with parafunctional habits

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Pink Esthetic Score (PES) | 6 months after delivery (18 months after IIP)
  The PES is based on seven parameters; mesial papilla, distal papilla, soft-tissue level, soft tissue contour, alveolar process deficiency, soft-tissue color, and texture. The peri-implant mucosa will be evaluated by the seven index points. The grading using the PES suggested by Fürhauser will be performed. The contralateral tooth and the adjacent soft tissue served as reference using a 0-1-2 scoring system, with 0 being the lowest and 2 being the highest value (Fürhauser et al., 2005).

SECONDARY OUTCOMES:
Bucco-palatal width | Before surgery - 12 months
  Measured with CBCT
Gingival thickness | Before surgery - 6 months - 12 months
  Measured with periodontal probe
Mid facial recession to assess the changes in tissue level | Before surgery - 3 months - 6 months - 9 months - 12 months
  Measured with 3D Viewer software
Interdental papillae height to assess changes in papilla height | Before surgery - 3 months - 6 months - 9 months - 12 months
  Measured with 3D Viewer software
Modified Plaque Index | 3 months - 6 months - 9 months - 12 months
  Measured with Periodontal probe
Modified Bleeding Index | 3 months - 6 months - 9 months - 12 months
  Measured with Periodontal probe
Patient satisfaction | 12 months
  Measured with Visual Analogue Scale (VAS). The patients will mark their satisfaction in a non-numerical 100 mm line ranging from "not at all satisfied=0" (left) to "very satisfied=100" (right), for each implant
Volumetric analysis of buccal contour to assess changes in buccal countour | Before surgery - 3 months - 6 months - 9 months - 12 months
  Measured with Extra oral scanning + 3D viewer software

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed I Abo El Futtouh, Master, Principal Investigator — Clinical Director of Implant Program - Misr International University; Khaled Abdel-Ghaffar, Professor, Study Director — Minister of Higher Education and Scientific Research; Inas S Hanna, Bsc, Study Director — Dentist/Researcher - IDCE; Nael A Mina, Bsc, Study Chair — Misr International University; Abdel Rahman A Abdel Rahman, Master, Study Chair — International Dental Contiuing Education; Ahmed F Mostafa, Bsc, Study Chair — International Dental Contiuing Education
Locations (2):
- Egypt (2):
  - International Dental Contining Education Centre (IDCE), Cairo
  - Misr International University, Cairo

IPD SHARING:
Plan to Share IPD: Yes
All data can be shared
Supporting Information: SAP, CSR
Time Frame: One year
Access Criteria: Principal investigator

REFERENCES:
- [Background] Gluckman H, Salama M, Du Toit J. Partial Extraction Therapies (PET) Part 2: Procedures and Technical Aspects. Int J Periodontics Restorative Dent. 2017 May/Jun;37(3):377-385. doi: 10.11607/prd.3111. PMID 28402349
- [Background] Fuentealba R, Jofre J. Esthetic failure in implant dentistry. Dent Clin North Am. 2015 Jan;59(1):227-46. doi: 10.1016/j.cden.2014.08.006. Epub 2014 Sep 26. PMID 25434568
- [Background] Esposito M, Grusovin MG, Felice P, Karatzopoulos G, Worthington HV, Coulthard P. The efficacy of horizontal and vertical bone augmentation procedures for dental implants - a Cochrane systematic review. Eur J Oral Implantol. 2009 Autumn;2(3):167-84. PMID 20467628
- [Background] Chen ST, Buser D. Esthetic outcomes following immediate and early implant placement in the anterior maxilla--a systematic review. Int J Oral Maxillofac Implants. 2014;29 Suppl:186-215. doi: 10.11607/jomi.2014suppl.g3.3. PMID 24660198
- [Background] Buser D, Martin W, Belser UC. Optimizing esthetics for implant restorations in the anterior maxilla: anatomic and surgical considerations. Int J Oral Maxillofac Implants. 2004;19 Suppl:43-61. PMID 15635945
- [Background] Grunder U, Gracis S, Capelli M. Influence of the 3-D bone-to-implant relationship on esthetics. Int J Periodontics Restorative Dent. 2005 Apr;25(2):113-9. PMID 15839587
- [Background] Araujo MG, Lindhe J. Dimensional ridge alterations following tooth extraction. An experimental study in the dog. J Clin Periodontol. 2005 Feb;32(2):212-8. doi: 10.1111/j.1600-051X.2005.00642.x. PMID 15691354
- [Background] Araujo MG, Sukekava F, Wennstrom JL, Lindhe J. Tissue modeling following implant placement in fresh extraction sockets. Clin Oral Implants Res. 2006 Dec;17(6):615-24. doi: 10.1111/j.1600-0501.2006.01317.x. PMID 17092218
- [Background] Chen ST, Buser D. Clinical and esthetic outcomes of implants placed in postextraction sites. Int J Oral Maxillofac Implants. 2009;24 Suppl:186-217. PMID 19885446
- [Background] Horvath A, Mardas N, Mezzomo LA, Needleman IG, Donos N. Alveolar ridge preservation. A systematic review. Clin Oral Investig. 2013 Mar;17(2):341-63. doi: 10.1007/s00784-012-0758-5. Epub 2012 Jul 20. PMID 22814758
- [Background] Masaki C, Nakamoto T, Mukaibo T, Kondo Y, Hosokawa R. Strategies for alveolar ridge reconstruction and preservation for implant therapy. J Prosthodont Res. 2015 Oct;59(4):220-8. doi: 10.1016/j.jpor.2015.04.005. Epub 2015 May 26. PMID 26022542
- [Background] De Risi V, Clementini M, Vittorini G, Mannocci A, De Sanctis M. Alveolar ridge preservation techniques: a systematic review and meta-analysis of histological and histomorphometrical data. Clin Oral Implants Res. 2015 Jan;26(1):50-68. doi: 10.1111/clr.12288. Epub 2013 Nov 1. PMID 27007188
- [Background] Luckerath W, Roder L, Enkling N. The Effect of Primary Stabilization of the Graft in a Combined Surgical and Prosthodontic Ridge Preservation Protocol: A Prospective Controlled Clinical Pilot Study. Int J Periodontics Restorative Dent. 2018 May/Jun;38(3):e49-e58. doi: 10.11607/prd.3172. PMID 29641631
- [Background] Kan JY, Rungcharassaeng K. Immediate placement and provisionalization of maxillary anterior single implants: a surgical and prosthodontic rationale. Pract Periodontics Aesthet Dent. 2000 Nov-Dec;12(9):817-24; quiz 826. PMID 11405020
- [Background] Kan JYK, Rungcharassaeng K, Deflorian M, Weinstein T, Wang HL, Testori T. Immediate implant placement and provisionalization of maxillary anterior single implants. Periodontol 2000. 2018 Jun;77(1):197-212. doi: 10.1111/prd.12212. Epub 2018 Feb 25. PMID 29478284
- [Background] Tarnow DP, Chu SJ, Salama MA, Stappert CF, Salama H, Garber DA, Sarnachiaro GO, Sarnachiaro E, Gotta SL, Saito H. Flapless postextraction socket implant placement in the esthetic zone: part 1. The effect of bone grafting and/or provisional restoration on facial-palatal ridge dimensional change-a retrospective cohort study. Int J Periodontics Restorative Dent. 2014 May-Jun;34(3):323-31. doi: 10.11607/prd.1821. PMID 24804283
- [Background] Chu SJ, Salama MA, Garber DA, Salama H, Sarnachiaro GO, Sarnachiaro E, Gotta SL, Reynolds MA, Saito H, Tarnow DP. Flapless Postextraction Socket Implant Placement, Part 2: The Effects of Bone Grafting and Provisional Restoration on Peri-implant Soft Tissue Height and Thickness- A Retrospective Study. Int J Periodontics Restorative Dent. 2015 Nov-Dec;35(6):803-9. doi: 10.11607/prd.2178. PMID 26509983
- [Background] Chu SJ, Saito H, Salama MA, Garber DA, Salama H, Sarnachiaro GO, Reynolds MA, Tarnow DP. Flapless Postextraction Socket Implant Placement, Part 3: The Effects of Bone Grafting and Provisional Restoration on Soft Tissue Color Change-A Retrospective Pilot Study. Int J Periodontics Restorative Dent. 2018 Jul/Aug;38(4):509-516. doi: 10.11607/prd.3571. PMID 29889914
- [Background] Akin R. A New Concept in Maintaining the Emergence Profile in Immediate Posterior Implant Placement: The Anatomic Harmony Abutment. J Oral Maxillofac Surg. 2016 Dec;74(12):2385-2392. doi: 10.1016/j.joms.2016.06.184. Epub 2016 Jul 1. PMID 27475245
- [Background] Janakievski J. Case Report : Maintenance of Gingival Form Following Immediate Implant Placement - The Custom-Healing Abutment. Adv Esthet Interdiscip Dent. 2007;3(4):4-7
- [Background] Mihali S. Maintaining Tissue Architecture in Immediate Implant Placement Following Extraction of Natural Teeth Using Custom Healing Screw. Biomed J Sci Tech Res. 2018
- [Background] Zuiderveld EG, Meijer HJA, den Hartog L, Vissink A, Raghoebar GM. Effect of connective tissue grafting on peri-implant tissue in single immediate implant sites: A RCT. J Clin Periodontol. 2018 Feb;45(2):253-264. doi: 10.1111/jcpe.12820. Epub 2017 Dec 5. PMID 28941303
- [Background] Kan JY, Rungcharassaeng K, Morimoto T, Lozada J. Facial gingival tissue stability after connective tissue graft with single immediate tooth replacement in the esthetic zone: consecutive case report. J Oral Maxillofac Surg. 2009 Nov;67(11 Suppl):40-8. doi: 10.1016/j.joms.2009.07.004. PMID 19835749
- [Background] Kolerman R, Nissan J, Mijiritsky E, Hamoudi N, Mangano C, Tal H. Esthetic assessment of immediately restored implants combined with GBR and free connective tissue graft. Clin Oral Implants Res. 2016 Nov;27(11):1414-1422. doi: 10.1111/clr.12755. Epub 2016 Jan 7. PMID 26743894